CLINICAL TRIAL: NCT05479318
Title: A Global Approach to Tackle Cognitive Decline
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The University of New South Wales (Other); University of Oxford (Other); University College, London (Other); Umeå University (Other); Max Planck Institute for Human Development (Other); National University of Singapore (Other)
Responsible Party: Principal Investigator, Bonnie Yin Ka LAM, Research Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2022.119
Record Dates: First submitted 2022-05-18; First posted 2022-07-29 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The number of people suffering from dementia in Asia (22.9 million) is more than twice the numbers in Europe (10.5 million) or the Americas (9.4 million), as recorded in the global impact of dementia in the World Alzheimer Report 2015.1 This dementia tsunami will continue to rise and the estimated number is 67 million in 2050 in Asia alone, which will be 2 to 3 times higher than the estimates for Europe (19 million) or the Americas (30 million). Devising and implementing preventive strategies against dementia is of paramount importance. The proposed project will be able to establish the associations between VRFs and cognition across cohorts with cultural, ethnical, and demographical variations. This study will generate data for evidence-based knowledge for globally implementable and effective preventive strategies for cognitive impairment and dementia.

DETAILED DESCRIPTION:
Participants will be retrospectively selected from a Hong Kong Chinese cohort, a Singaporean cohort, a British cohort, two European cohorts, and an Australian cohort.

Subjects from the above listed cohorts who fit the study criteria will be selected for this study.

Demographical information, clinical, vascular risk factors, MRI images and cognitive data will be retrieved from the cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly community-dwelling individuals aged over 60 years old;
2. those with at least 2 time points of detailed cognitive measurements, with 2-3 years of assessment interval;
3. with at least 1 timepoint of MRI (T1, FLAIR, and DTI).

Exclusion Criteria:

1. subjects with stroke, dementia, and other neurological diseases at baseline;
2. those without longitudinal cognitive data;
3. those without MRI data available.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be retrospectively selected from 7 cohorts from Hong Kong, Australia, Singapore and Europe areas.
Sampling Method: Non-Probability Sample
Enrollment: 1502 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Record of any vascular risk factors | Baseline
  medical history of hypertension, diabetes mellitus, hyperlipidemia, smoking and drinking, record unit as yes or no
Record of triglyceride level | Baseline
  triglyceride level, as one of vascular risk factors, unit as mmol/L
Record of high-density-lipoprotein level, | Baseline
  high-density-lipoprotein level, as one of the vascular risk factors, unit as mmol/L
Record of low-density-lipoprotein level, | Baseline
  low-density-lipoprotein level, as one of the vascular risk factors, unit as mmol/L
Record of total cholesterol level, | Baseline
  total cholesterol level, as one of the vascular risk factors, unit as mmol/L
Record of glycated hemoglobin | Baseline
  glycated hemoglobin, as one of the vascular risk factors, unit as percentage
Record of fasting blood glucose | Baseline
  fasting blood glucose from blood results, as one of vascular risk factors, unit as mmol/L
Record of blood pressure | Baseline
  Blood pressure, as one of vascular risk factors, unit as mmHg
Record of pulse | Baseline
  Pulse rate, as one of vascular risk factors, unit as bpm
Change of Mini-Mental State Examination | Baseline and 3rd year follow up
  Mini-Mental State Examination is used for measuring general cognition including the domains of attention and processing speed, executive function, memory, visuospatial function, and animal fluency.
Change of Montreal Cognitive Assessment | Baseline, 1 yr, 2yr and 3rd year follow ups
  Montreal Cognitive Assessment is used for measuring general cognition including the domains of attention and processing speed, executive function, memory, visuospatial function, and animal fluency.
Changes of brain white matter abnormalities | Baseline and 1 yr, 2yr and 3rd year follow ups
  brain white matter abnormalities can be observed through the FLAIR sequence of brain MRI images

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Yin Ka Lam, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, N.T., Hong Kong

IPD SHARING:
Plan to Share IPD: No